CLINICAL TRIAL: NCT05665114
Title: Clinical Study on the Safety and Efficacy of QN-030a in Acute Myeloid Leukemia
Brief Title: Natural Killer(NK) Cell Therapy in r/r AML
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Qihan Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Dr., Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QN030aAL
Record Dates: First submitted 2022-12-13; First posted 2022-12-27 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; fludarabine; Cytarabine; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QN-030a (Experimental): QN-030a in Adult subjects with r/r AML
  Interventions: Drug: QN-030a; Drug: Cyclophosphamid; Drug: Fludarabine; Drug: Cytarabine; Drug: VP-16

INTERVENTIONS:
Drug: QN-030a — NK cell therapy
Drug: Cyclophosphamid — Lympho-conditioning Agent
Drug: Fludarabine — Lympho-conditioning Agent
Drug: Cytarabine — Lympho-conditioning Agent
Drug: VP-16 — Lympho-conditioning Agent

SUMMARY:
This is an open-label, Phase I study of QN-030a (allogeneic NK cell therapy) in relapse/refractory Acute Myeloid Leukemia (AML).

This clinical study is to evaluate the safety, tolerability and preliminary efficacy of QN-030a in patients with r/r AML, where a "3+3" enrollment schema will be utilized at dose escalation stage. Up to 18 patients will be enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of signed and dated informed consent form (ICF)
* ≥18 years old
* Diagnosis of r/r AML
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Adequate organ function as defined in the protocol
* Donor specific antibody (DSA) to QN-030a: MFI <= 2000

Key Exclusion Criteria:

* Allergic to drug used in this study
* Accept other anti-tumor drugs/therapies within certain time of day 0 (first QN-030a dose infusion), time window and drug defined in the protocol.
* received systemic immunosuppressive therapy within 7 days of day 0, or likely to require systemic immunosuppressive therapy
* Acute Promyelocytic Leukemia (APL)
* Central nervous system Leukemia.
* Uncontrolled, active clinically significant infection
* Clinically significant cardiovascular disease as defined in the protocol
* Known HIV infection, active Hepatitis B (HBV) or Hepatitis C (HCV) infection
* History of central nervous system (CNS) disease such as stroke, epilepsy.
* Females are pregnant or lactating
* Investigator-assessed presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-12-24 (Estimated); Primary Completion 2023-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to approximately 2 years after last dose of QN-030a
Incidence of dose adjustment or discontinuation due to NK cell toxicities | Up to approximately 2 years after last dose of QN-030a
Incidence of subjects with Dose Limiting Toxicities within each dose level cohort | 28 Days from first dose of QN-030a
Determine the Maximum tolerated dose (MTD) and RP2D | 28 Days from first dose of QN-030a

SECONDARY OUTCOMES:
Overall Response Rate(ORR) of QN-030a in r/r AML | Up to approximately 2 years after last dose of QN-030a
  Proportion of subjects who achieve a CR, CRi, CRMRD-, MLFS, or PR, as determined by investigator.
Relapse-free survival (RFS) of QN-030a in r/r AML | Up to approximately 2 years after last dose of QN-030a
Time to Response (TTR) of QN-030a in r/r AML | Up to approximately 2 years after last dose of QN-030a
Event-free survival (EFS) of QN-030a in r/r AML | Up to approximately 2 years after last dose of QN-030a
Overall Survival (OS) of QN-030a in r/r AML | Up to approximately 2 years after last dose of QN-030a
Determination of the pharmacokinetics (PK) of QN-030a cells in peripheral blood | Up to approximately 2 years after last dose of QN-030a
  The PK of QN-030a in peripheral blood will be reported as the relative percentage of product (QN-030a) DNA versus patient DNA (% chimerism) measured from blood samples at the specified time points
Evaluate the immunogenicity features of QN-030a | Up to approximately 2 years after last dose of QN-030a
  The Donor specific antibody (DSA) and T cell receptor (TCR) will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China